CLINICAL TRIAL: NCT03142880
Title: Spinal Ropivacaine for Cesarean Delivery: A Comparison of Commonly Hyperbaric and Marginally Hyperbaric Solutions
Brief Title: Spinal Marginally Hyperbaric Ropivacaine for Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZX01
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia, Spinal
Keywords: marginally hyperbaric; ropivacaine; cesarean

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- commonly hyperbaric ropivacaine group (Active Comparator): This group will receive spinal anesthesia with commonly hyperbaric ropivacaine solution,which was made by adding 50% glucose to the plain ropivacaine commercially availablethe to make it's density is close to commonly hyperbaric bupivacaine.
  Interventions: Combination Product: hyperbaric ropivacaine
- marginally hyperbaric ropivacaine group (Experimental): This group will receive spinal anesthesia with marginally hyperbaric ropivacaine,which was made by adding 5% glucose to the plain ropivacaine commercially availablethe to make it's density is slightly denser than cerebrospinal fluid but much less denser than commonly hyperbaric bupivacaine/ropivacaine.
  Interventions: Combination Product: hyperbaric ropivacaine

INTERVENTIONS:
Combination Product: hyperbaric ropivacaine — We change the density of ropivacaine solution to make it into an marginally hyperbaric state or into an commonly hyperbaric state.and we hypothesized that the marginally hyperbaric ropivacaine will get a similar efficacy to commonly hyperbaric solutions but a more steadily hemodynamic status.
  Other Names: commonly or marginally hyperbaric ropivacaine

SUMMARY:
BACKGROUND: One previous study has confirmed that the marginally hyperbaric solutions of bupivacaine can maintain good quality of anesthesia and get a more steadily hemodynamic status than commonly hyperbaric solutions, some authors confirmed the plain ropivacaine for cesarean section have a higher failure rate and commonly hyperbaric solutions of ropivacaine have a higher incidence of side reaction. It is unclear what the efficacy of spinal marginally hyperbaric ropivacaine for elective cesarean delivery.We hypothesized that the marginally hyperbaric ropivacaine will get a similar efficacy to commonly hyperbaric solutions but a more steadily hemodynamic status.

OBJECTIVE In this prospective, randomized, double-blinded study, Investigator will compare the clinical efficacy and adverse effect of spinal anesthesia with commonly hyperbaric and marginally hyperbaric ropivacaine for elective cesarean delivery.

Main outcome measures: The maximum cephalad sensory block level; the change of continuous cerebral oxygen desaturation (ScO2) over time; the incidence of hypotension and nausea and vomiting; the change of invasive arterial pressure; the consumption of ephedrine; the incidence of shivering; the onset time to T8 dermatome; the quality of anesthesia (efficacy of motor block and sensory block)

DETAILED DESCRIPTION:
INTRODUCTION:

One previous study has confirmed that the marginally hyperbaric solutions of bupivacaine can maintain good quality of anesthesia and get a more steadily hemodynamic status than commonly hyperbaric solutions, some authors confirmed the plain ropivacaine for cesarean section have a higher failure rate and commonly hyperbaric solutions of ropivacaine have a higher incidence of side reaction such as hypotension. It is unclear what the efficacy of spinal marginally hyperbaric ropivacaine for elective cesarean delivery.The investigator of this study hypothesized that the marginally hyperbaric ropivacaine would get a similar efficacy to commonly hyperbaric solutions but a more steadily hemodynamic status.In this prospective, randomized, double-blinded study, Investigator will compare the clinical efficacy and adverse effect of spinal anesthesia with commonly hyperbaric and marginally hyperbaric ropivacaine for elective cesarean delivery.

Ethical approval for this clinical trial (Ethical Committee No.) was provided by the Ethics Committee of Qilu Hospital of Shandong University (Qingdao), Qingdao, China on 1 February 2016. Informed written consent will be obtained from all patients. Investigator expected to recruit 120 Pregnant women who will scheduled for elective cesarean section and meet the inclusion criteria.

A computer-generated random number sequence will be used for group allocation. To ensure the study will be double blinded, the anesthesiologist who will administer the anesthesia will take no other part in the study, whilst another anesthesiologist blind to the allocation will collected intraoperative and postoperative data. The patients would be unaware of the treatment allocation. Women will be randomised into two groups: the commonly hyperbaric group (CH) will receive ropivacaine solution with 8.3% glucose; group marginally hyperbaric group (MH) will receive ropivacaine solution with 0.83% glucose; Density will be determined by using a digital density meter (DMA4500M; Anton Paar GmbH, Graz, Austria) at 37°C.Fifteen minutes prior to administration of anesthesia, the ropivacaine solution will be prepared by one nurse who is blind to the patient allocation.Commomly hyperbaric ropivacaine solutions will be made of 0.75% ropivacaine + 50% glucose + isotonic saline and Marginally hyperbaric solutions will be made of 0.75% ropivacaine +5% glucose + isotonic saline. The doses of ropivacaine and the volume of spinal solution will be same and only the density of the solution will be different.

When the patient arrived at the operating room, an IV cannula will be inserted in one forearm. Standard monitoring with electrocardiography and pulse oximetry and cerebral oxygen saturation(ScO2) and invasive blood pressure (IBP) will be attached.

During the operation, the room temperature will be kept at 24°C. The body temperature of each patient will be maintained by an electric warming blanket and infusion heating device.

The data of systolic pressure and ScO2 wil be recorded at 5-6 second intervals on the device's accessory disk drive for later analysis. To establish a baseline for blood pressure and ScO2. No prehydration will be given. Lactated Ringers' solution at 0.4 ml kg-1 min-1 will be infused after anesthesia. Supplemental oxygen is planned to be administered in case SpO2 values would be below 91%.

The combined spinal-epidural anesthesia (CSEA) would be performed in the lateral position at the intervertebral space between L3 and L4. Then, spinal solution will be injected intrathecalley after CSF releas. The epidural catheter will be inserted. The patient will be immediately placed in a supine position with 15° left tilt. Completion of the spinal injection would be considered as time zero. The sensory block will be determined by pinprick along both sides of the midclavicular line at 2 min intervals post injection. The sensory block had not reached T8 before surgery, or there was moderate pain during the skin incision, spinal anesthesia would be considered to have failed.

The efficacy of anesthesia would be evaluated using three criteria: lower limb motor block, muscle relaxation and pain during skin incision and abdominal exploration.

To treat intraoperative hypotension, 6mg ephedrine will be injected followed by 3 mg every 2 min until the blood pressure was restored to normal. Instances of nausea, vomiting, shivering and pruritus will be also recorded.

After delivery, Apgar scores will be assessed at 1 and 5 min by the attending pediatrician.

On the basis of the results of a pilot study, 40 patients in each group were needed to compare a two-segment difference in the upper sensory level and 30 % difference in the incidence of hypotension at a significance level of P less than 0.05 with 80% power. However, We expect to enroll 120 patients to get a more precise result.

For IBP and ScO2 the median value of the sliding averages of the 30-second period before spinal induction will be used as the baseline value for the figures and statistical analyses. Time 0 for hemodynamic analyses will be defined as the end of spinal injection. This two variables analyses will be run for the first 15 minutes, which almost equaled to the interval from induction of spinal anesthesia to delivery.

SPSS 16.0 will be used for data analysis. T-test would be used to assess the difference in sensory block level amongst the groups, The linear mixed model to analyze the continuous changes in systolic pressure and ScO2 over time. X2 test for trends would be used to test the association between adverse effects of anesthesia and the groups. In all cases, a P value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were scheduled for elective caesarean section and met the criteria for the American Society of Anesthesiologists (ASA) physical status classes 1 to 2 were enrolled in this study. Inclusion criteria were age between 20 and 42 years, height between 160 and 180 cm.

Exclusion Criteria:

* They had dysfunctional coagulation; had pregnancy-induced hypertension; or had infection around the anesthesia puncture site; or multiple pregnancies, suspected fetal abnormality, and if the gestational age of the infant was less than 36 weeks.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The maximum cephalad sensory block level | During 50 min post spinal injection
  The highest cephalad sensory block level is determined by pinprick along both sides of the midclavicular line.

SECONDARY OUTCOMES:
The incidence of hypotension | During 50 min post spinal injection
  The systolic pressure <80% of baseline value or<90 mm Hg
The change rate of invasive arterial pressure | During 15 min post spinal injection
  The invasive arterial pressure decline rate over time after spinal anesthesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang WX, Li JJ, Bu HM, Fu ZJ. Spinal anaesthesia with low-dose bupivacaine in marginally hyperbaric solutions for caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jul;32(7):493-8. doi: 10.1097/EJA.0000000000000112. PMID 25032943
- [Background] Khaw KS, Ngan Kee WD, Wong M, Ng F, Lee A. Spinal ropivacaine for cesarean delivery: a comparison of hyperbaric and plain solutions. Anesth Analg. 2002 Mar;94(3):680-5; table of contents. doi: 10.1097/00000539-200203000-00037. PMID 11867397